CLINICAL TRIAL: NCT00789009
Title: Clinical and Immunologic Monitoring of Patients With Known or Suspected HIV Infection
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090030; 09-I-0030
Record Dates: First submitted 2008-11-08; First posted 2008-11-11 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-11-26

CONDITIONS: HIV
Keywords: Opportunistic Infections; AIDS; Natural History
MeSH Terms: conditions — Opportunistic Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Consist of HIV positive patients recruited from the Washington DC metropolitan area who will receive long-term care for their HIV infection through the NIAID/CCMD HIV clinic
- Group 2: Patients with known or suspected HIV infection, referred to a NIAID/CCMD investigator for reasons such as testing to diagnose or exclude HIV disease or assistance with HIV-related problems.

SUMMARY:
This study will investigate HIV infection and associated conditions by monitoring infected patients. The study will also serve as a means for recruiting HIV-infected individuals to NIAIDs ongoing clinical and laboratory studies and supporting the institute s infectious disease training program by providing Infectious Disease fellows with ongoing training in the management of HIV infection.

People 18 years of age and older with suspected or confirmed HIV infection who live in the Washington, D.C., metropolitan area may be eligible for this study. Physician referral is required.

Participants come to the NIH Clinical Center a minimum of once every 3 to 4 months for evaluation with a physical examination; blood tests for research purposes, safety, immune status and viral load; and response to any treatment they may be receiving. Other procedures, such as a biopsy, are done only as needed for standard medical practice, and informed consent is obtained before any such procedure is done. Treatment offered is consistent with standard medical practice; no experimental treatments are offered under this protocol.

DETAILED DESCRIPTION:
This study is designed as a prospective natural history study with ongoing monitoring of HIV infection and HIV-related disease processes. The overall protocol Objective is to determine the long-term clinical outcome of treated HIV infection and investigate aspects of the host immune response that may predict outcomes. Minimal studies scheduled for each visit include: monitoring of immune status and viral load, routine safety laboratory tests, and collection of blood for research and storage. Medical treatment of HIV infection will be provided in accordance with standard medical practice. Specific HIV treatment regimens will be in accordance with standard medical practice and not constitute research.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients are subject to selection by the Principal Investigator, and will satisfy all of the following inclusion criteria:

1. HIV-infection as documented by positive HIV ELISA and Western Blot or positive assay for HIV RNA (serum or plasma). Patients may also be included if they have laboratory or clinical evidence suggestive of possible HIV-infection.
2. Age 18 years or older.
3. Ability and willingness of subject to understand study requirements and give written informed consent.
4. Group I patients are required to have a primary care provider outside NIH to manage non-HIV medical problems. Group II patients must have a referring physician or clinic that will continue to manage HIV and non-HIV medical care.
5. For Group I patients, residence within the greater Washington DC area (approximately within a 100-mile radius of the NIH Bethesda campus) is required.

EXCLUSION CRITERIA:

A prospective study subject will be ineligible for this study if he or she satisfies either of the following criteria:

1. Has active drug or alcohol use or dependence or any other condition that, in the opinion of the investigator, would interfere with adherence to study requirements.
2. Refuses to allow collection and storage of samples for research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The first subgroup will consist of patients recruited from the Washington DC metropolitan area who will receive long-term care for their HIV infection through the NIAID/CCMD HIV clinic. The second subgroup will consist of patients with known or suspected HIV infection who have been referred to a NIAID/CCMD investigator for reasons such as further testing to diagnose or exclude HIV disease, assistance with the diagnosis or management of acute HIV-related problems. This latter subgroup of patients will be followed on a short-term (12 months or less). Following discharge from the protocol, Group II patients will be returned to the care of their referring physicians.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2008-11-20 (Actual)

PRIMARY OUTCOMES:
This study will provide a clinically well-characterized cohort of HIV infected individuals to support ongoing clinical and laboratory based NIAID intramural research programs described above. | Every 3 to 6 months
  Laboratory results and clinical data

SECONDARY OUTCOMES:
This study will support the NIAID Infectious Disease training program by providing fellows with ongoing training in the management of HIV infection. | Yearly
  Training

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Sneller, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aberg JA, Gallant JE, Anderson J, Oleske JM, Libman H, Currier JS, Stone VE, Kaplan JE; HIV Medicine Association of the Infectious Diseases Society of America. Primary care guidelines for the management of persons infected with human immunodeficiency virus: recommendations of the HIV Medicine Association of the Infectious Diseases Society of America. Clin Infect Dis. 2004 Sep 1;39(5):609-29. doi: 10.1086/423390. Epub 2004 Aug 11. No abstract available. PMID 15356773
- [Background] Dube MP, Stein JH, Aberg JA, Fichtenbaum CJ, Gerber JG, Tashima KT, Henry WK, Currier JS, Sprecher D, Glesby MJ; Adult AIDS Clinical Trials Group Cardiovascular Subcommittee; HIV Medical Association of the Infectious Disease Society of America. Guidelines for the evaluation and management of dyslipidemia in human immunodeficiency virus (HIV)-infected adults receiving antiretroviral therapy: recommendations of the HIV Medical Association of the Infectious Disease Society of America and the Adult AIDS Clinical Trials Group. Clin Infect Dis. 2003 Sep 1;37(5):613-27. doi: 10.1086/378131. Epub 2003 Aug 15. No abstract available. PMID 12942391
- [Background] Le Saout C, Hasley RB, Imamichi H, Tcheung L, Hu Z, Luckey MA, Park JH, Durum SK, Smith M, Rupert AW, Sneller MC, Lane HC, Catalfamo M. Chronic exposure to type-I IFN under lymphopenic conditions alters CD4 T cell homeostasis. PLoS Pathog. 2014 Mar 6;10(3):e1003976. doi: 10.1371/journal.ppat.1003976. eCollection 2014 Mar. PMID 24603698
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2009-I-0030.html